CLINICAL TRIAL: NCT03556878
Title: Implementing and Sustaining a Transdiagnostic Sleep and Circadian Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adapted_MH105513
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Sleep Disorders, Circadian Rhythm; Sleep Disorder; Acceptability; Feasibility; Adaptation; Implementation Research
Keywords: Circadian rhythm disorders; Sleep disorders; Acceptability; Adaptation; Feasibility
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Sleep Wake Disorders; Chronobiology Disorders

STUDY DESIGN:
Intervention Model Description: This is a 'treatment development' pilot study in which we intended to continue to develop and adapted 'Fitted TranS-C' as we gain experience. At the outset of the study, it involves 4 x 20-30 minute sessions. It utilizes four cross-cutting, 3 core and 1 optional modules from Standard TranS-C. All participants will get the same Fitted Trans-C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fitted TranS-C (Experimental): Fitted TranS-C involves 4 x 20-30 minute sessions. It involves selected cross-cutting, core and optional modules from Standard TranS-C.
  Interventions: Behavioral: Fitted Transdiagnostic Sleep and Circadian intervention

INTERVENTIONS:
Behavioral: Fitted Transdiagnostic Sleep and Circadian intervention — Fitted TranS-C is an adapted version is designed to improve the fit with community needs and resources.
  Other Names: Fitted TranS-C

SUMMARY:
The goal is to collect pilot data on an adapted version of the Transdiagnostic Sleep and Circadian intervention (TranS-C), referred to as 'Fitted TranS-C'.

DETAILED DESCRIPTION:
Mental illness is often severe, chronic and difficult to treat. The sleep disturbance commonly experienced by individuals with a severe mental illness reduces capacity to function and contributes to key symptoms. This study seeks to collect pilot data on an adapted version of the Transdiagnostic Sleep and Circadian intervention (TranS-C). The adapted version will be referred to as 'Fitted TranS-C' as it is designed to improve the fit to delivery within community mental health centers. 'Fitted' treatments are needed because the context for implementation (community setting) typically differs from the original testing context (university setting) causing a lack of 'fit' between the setting and evidence based treatments.

ELIGIBILITY:
Inclusion Criteria:

* Can understand treatment in English
* Is not currently at risk for suicide or homicide
* Has not worked the night shift more than 2 nights per week in the past 3 months
* Is not pregnant or nursing
* Has a guaranteed bed to sleep in for the next month, which is not a shelter.

Exclusion Criteria:

* At risk for suicide or homicide
* Has worked the night shift more than 2 nights per week in the past 3 months
* Is pregnant or nursing
* Does not have a guaranteed bed to sleep in for the next month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
The acceptability of the intervention to providers will be assessed by the 'Acceptability of Intervention Measure' (AIM) | 4 weeks (i.e. post-treatment assessment)
  The AIM is a measure of the extent to which the intervention is acceptable to providers. The AIM is comprised of 4 questions rated on a 1 'completely disagree' to 5 'completely agree' scale. The responses to all four qus will be reported along with the summed total score.
PROMIS--Sleep Disturbance (PROMIS = Patient-Reported Outcomes Information System) | Pre-treatment and 4 weeks later (i.e. post-treatment assessment)
  Assesses sleep disturbance experienced by patients
CEQ (Treatment Evaluation Questionnaire) | 4 weeks (i.e. post-treatment assessment)
  Assesses patients' expectations of the treatment.

SECONDARY OUTCOMES:
Process evaluation/qualitative interview | 4 weeks (i.e. post-treatment assessment)
  Assessing the clients' and therapists' opinions of the treatment
MINI | Baseline only
  Index of psychiatric disorders

OTHER OUTCOMES:
Referral form | Baseline only
  Assesses participant suitability for the study

CONTACTS AND LOCATIONS:
Overall Officials: Allison G Harvey, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- UC Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No